CLINICAL TRIAL: NCT00553345
Title: Bladder Cancer Prognosis Programme (Incorporating SELENIB Trial) [TREATMENT]
Brief Title: Selenium and Vitamin E in Preventing Cancer Progression and Recurrence in Patients With Early-Stage Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000574080; CRUK-BCPP-2005-01-TREATMENT; ISRCTN13889738; EU-20768
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2010-02

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage 0 bladder cancer; stage I bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Selenium; Vitamin E; Chemoprevention

INTERVENTIONS:
Drug: selenium
Drug: vitamin E
Procedure: chemoprevention

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of selenium and vitamin E may stop cancer from growing or coming back.

PURPOSE: This randomized phase III trial is studying giving selenium together with vitamin E to see how well it works compared with a placebo in preventing cancer progression and recurrence in patients with early-stage bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate whether selenium and/or vitamin E (α-tocopherol) supplementation reduces the risk of recurrence and progression.

OUTLINE: This is a multicenter study. Patients are stratified by recurrence risk group (high vs intermediate) and treatment center and randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral selenium tablet and oral vitamin E capsule once daily.
* Arm II: Patients receive oral selenium tablet and oral placebo capsule once daily.
* Arm III: Patients receive oral placebo tablet and oral vitamin E capsule once daily.
* Arm IV: Patients receive oral placebo tablet and oral placebo capsule once daily.

In all arms, treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed every 6 months for 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologically confirmed non-muscle-invasive transitional cell carcinoma (< pT2)

  * Newly diagnosed disease
* Able to be randomized within twelve months of diagnostic transurethral resection bladder tumor/biopsy
* Must meet 1 of the following recurrence risk criteria:

  * Intermediate risk

    * Multiple G1 pTa (> 1)
    * Solitary G1 pTa (≥ 3 cm)
    * G2 pTa
    * G1 pT1
    * G2 pT1 (1 or 2 tumors)
  * High risk

    * G3 pTa
    * G3 pT1
    * Cis
    * Multiple G2 pT1 (3 or more foci)
  * Low risk

    * Solitary G1 pTa < 3 cm

PATIENT CHARACTERISTICS:

* Not pregnant or breast feeding
* No HIV infection
* No condition that, in the opinion of the local investigator, might interfere with the safety of the patient or evaluation of the trial objectives

PRIOR CONCURRENT THERAPY:

* No concurrent immunosuppressive therapy after organ transplantation
* No concurrent cyclosporine
* Those who currently use or have used selenium and/or vitamin E supplements will not be excluded, however, they must agree not to take supplements containing selenium and vitamin E above a pre-specified dosage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515
Dates: Start 2005-12

PRIMARY OUTCOMES:
Recurrence-free interval

SECONDARY OUTCOMES:
Overall survival time
Incidence of transitional cell carcinoma outside the bladder
Incidence of all other malignancies clinically diagnosed
Incidence of cardiovascular events
Quality of life as assessed at each follow-up visit by the quality of life instruments EORTC QLQ-C30, QLQ-BLS24 and QLQ-BLM30
Progression-free interval

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Zeegers, Study Chair — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, England, United Kingdom